CLINICAL TRIAL: NCT04464759
Title: LIMIT Melanoma: (Lysosomal Inhibition + Melanoma ImmunoTherapy) A Phase 1/2 Open Label Trial of Nivolumab and Hydroxychloroquine or Nivolumab/Ipilimumab and Hydroxychloroquine in Patients With Advanced Melanoma
Brief Title: A Study of Nivolumab and Hydroxychloroquine or Nivolumab/Ipilimumab and Hydroxychloroquine in Advanced Melanoma
Acronym: LIMIT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ravi Amaravadi, MD (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Ravi Amaravadi, MD, Associate Professor of Medicine, Abramson Cancer Center at Penn Medicine
Organization: Abramson Cancer Center at Penn Medicine (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 01620; IRB#835033 (Other: University of Pennsylvania)
Record Dates: First submitted 2020-06-08; First posted 2020-07-09 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Hydroxychloroquine; Ipilimumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 1a: Nivolumab and Hydroxychloroquine (HCQ) (Experimental): Dose escalation:
  Dose Level 1: HCQ 400 mg orally every 12 hours and nivolumab 480 mg IV every 4 weeks
  Dose Level 2: HCQ 600 mg orally every 12 hours and nivolumab 480 mg IV every 4 weeks
  Continue protocol treatment for up to 24 months until disease progression, unacceptable toxicity, withdrawal of consent, or other protocol-mandated study removal.
  Interventions: Drug: Nivolumab; Drug: Hydroxychloroquine
- Phase 2: Nivolumab and Hydroxychloroquine (HCQ) (Experimental): HCQ 400-600 mg (maximum tolerated dose from Phase 1a) orally every 12 hours and nivolumab 480 mg IV every 4 weeks
  Continue protocol treatment for up to 24 months until disease progression, unacceptable toxicity, withdrawal of consent, or other protocol-mandated study removal.
  Interventions: Drug: Nivolumab; Drug: Hydroxychloroquine
- Phase 1b: Nivolumab + Ipilimumab +Hydroxychloroquine (HCQ) (Experimental): HCQ 400-600 mg orally every 12 hours and nivolumab 3 mg/kg IV plus ipilimumab 1 mg/kg IV every 3 weeks x4 cycles
  Then 6 weeks after the last dose of ipilimumab/nivolumab begin maintenance nivolumab 480 mg IV every 4 weeks
  Continue protocol treatment for up to 24 months until disease progression, unacceptable toxicity, withdrawal of consent, or other protocol-mandated study removal.
  Interventions: Drug: Nivolumab; Drug: Hydroxychloroquine; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Combination of nivolumab and hydroxychloroquine OR nivolumab, hydroxychloroquine and ipilimumab
  Other Names: Opdivo®
Drug: Hydroxychloroquine — Combination of nivolumab and hydroxychloroquine OR nivolumab, hydroxychloroquine and ipilimumab
  Other Names: Plaquenil
Drug: Ipilimumab — Combination of nivolumab, hydroxychloroquine and ipilimumab
  Other Names: YERVOY®
  Arms: Phase 1b: Nivolumab + Ipilimumab +Hydroxychloroquine (HCQ)

SUMMARY:
This study will evaluate the safety, tolerability and efficacy (objective response rate) of using hydroxychloroquine (HCQ) in combination with nivolumab and ipilimumab or with nivolumab alone in subjects with advanced/metastatic melanoma.

DETAILED DESCRIPTION:
There are three parts to this Phase 1/2 study in subjects with advanced melanoma:

Phase 1a will identify the MTD and preliminary safety of combination hydroxychloroquine and nivolumab therapy.

Phase 1b will identify the MTD and preliminary safety of hydroxychloroquine administered in conjunction with nivolumab and ipilimumab therapy

Phase 2 will assess the clinical efficacy of combination hydroxychloroquine and nivolumab therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological evidence of melanoma, unresectable Stage III or Stage IV, any genotype, and any programmed death-ligand 1 (PD-L1) immunohistochemistry (IHC) status
* Phase 1a: nivolumab + HCQ: any prior treatment, or treatment naïve
* Phase 2: nivolumab + HCQ:
* - - Cohort 2a: prior immunotherapy in the adjuvant or metastatic setting is required
* - - Cohort 2b: anti-PD-1 Ab-naïve, but may have received any prior other therapy
* Phase 1b nivolumab + ipilimumab + HCQ: anti-PD-1 refractory
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* At least one measurable site of disease by RECIST 1.1 criteria that has not been previously irradiated.
* Fresh or archived primary or metastatic tissue available for submission for correlative analyses
* Negative serum pregnancy test within 28 days prior to commencement of dosing in premenopausal women. Negative urine pregnancy test within 24 hours of starting treatment.
* Able to swallow and retain oral medication and no clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* Adequate baseline organ function

Exclusion Criteria:

* Known serious concurrent infection or medical illness, including psychiatric disorders, which would jeopardize the ability to receive the protocol treatment with reasonable safety.
* Pregnant or breast-feeding.
* Patients with brain metastases treated with whole brain radiation that have been stable for 2 months are eligible; patients with brain metastases treated with gamma knife or surgery are allowed to participate after 2 weeks have elapsed since their procedure. Subjects are excluded if they have leptomeningeal disease or metastases causing spinal cord compression that are symptomatic or untreated or not stable for greater than or equal to 3 months (documented by imaging) or requiring corticosteroids greater than 20 mg prednisone equivalent daily.
* Must have discontinued active immunotherapy, chemotherapy, or investigational anticancer therapy at least 4 weeks prior to entering the study and oral targeted therapy at least 2 weeks prior to entering the study.
* All prior anti-cancer treatment-related toxicities (except alopecia and laboratory values listed in protocol eligibility) must be less than or equal to Grade 1 or irreversible (hypophysitis) according to the Common Terminology Criteria for Adverse Events version 5 at the time of starting treatment. Patients that are asymptomatic on low dose maintenance hormone replacement delivered at a stable dose for prior toxicities are eligible.
* Prior or concurrent cancer therapy. Active immunotherapy, chemotherapy, or investigational anticancer therapy within 4 weeks prior to entering the study or oral targeted therapy within 2 weeks prior to entering the study
* Phase 2 nivolumab + HCQ Cohort B: No prior immunotherapy is permitted
* Patients known to be experiencing an objective partial response to immunotherapy at the time of study enrollment.
* History of malignancy other than disease under study within 3 years of study enrollment EXCEPT: history of completely resected non-melanoma skin cancer, or history of indolent second malignancies are eligible.
* Diagnosis of severe autoimmune disease requiring immunosuppressive medications. Patients with adrenal insufficiency on replacement dose steroids are eligible.
* History of interstitial lung disease or chronic pneumonitis unrelated to prior immunotherapy. Prior interstitial pneumonitis related to immunotherapy that was completely treated with no need for ongoing clinical management is allowed.
* Due to risk of disease exacerbation patients with porphyria or psoriasis are ineligible unless the disease is well controlled and they are under the care of a specialist for the disorder who agrees to monitor the patient for exacerbations.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to study drug, or excipients or to dimethyl sulfoxide.
* Patients receiving cytochrome P450 enzyme-inducing anticonvulsant drugs (i.e. phenytoin, carbamazepine, Phenobarbital, primidone or oxcarbazepine) within 4 weeks of the start of the study treatment
* Current use of a prohibited medication as described in section on Potential for Drug-Drug Interaction.
* History or evidence of increased cardiovascular risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2020-10-21 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Maximum tolerated dose (MTD) - Number of Subjects with Dose-limiting Toxicities | From first dose of protocol treatment to 16 to 32 weeks
  To determine the MTD and preliminary safety of HCQ when administered in conjunction with one of the following treatments in patients with advanced melanoma:
  * HCQ administered in combination with nivolumab; or
  * HCQ administered in combination with nivolumab and ipilimumab followed by maintenance nivolumab
Phase 2: Objective Response Rate (ORR) | 12 months
  To assess the ORR as measured by RECIST v1.1. in subjects with advanced melanoma

SECONDARY OUTCOMES:
Progression-free survival | From start of treatment to first progression, death due to any cause or last patient contact alive and progression-free over 24 months
  The time from protocol treatment start to disease progression, death due to any cause, or last contact alive and progression-free over 24 months
1 year survival rate | From start of treatment to one year
  Percentage of subjects alive at one year from start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Amaravadi, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center at University of Pennsylvania, Philadelphia, Pennsylvania, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/59/NCT04464759/Prot_SAP_000.pdf